CLINICAL TRIAL: NCT06793865
Title: Effect of Russian Current Stimulation for Anterior Tibial Group on Postural Stability and Risk of Falling in Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Refaat Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005504
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Russian Current Stimulation + selected physical therapy exercise (Experimental): Patients received Russian current stimulation for 20 minutes and physical therapy for 40 minutes, 3 times/week for 6 weeks.
  Interventions: Other: Russian Current Stimulation for Anterior Tibial Group; Other: Selected physical therapy exercise for both limbs
- Placebo Russian Current Stimulation + selected physical therapy exercise (Placebo Comparator): All patients in this group received Russian current for 20 minutes as placebo in addition to the same selected physical therapy exercise for both limbs for 40 minutes.
  Interventions: Other: Placebo Russian Current Stimulation for Anterior Tibial Group; Other: Selected physical therapy exercise for both limbs

INTERVENTIONS:
Other: Russian Current Stimulation for Anterior Tibial Group — Parameters were adjusted as the following frequency of 2.5 kHz and 50 bursts per second with 50 pulses per burst. The stimulus was applied for a 10 seconds "on" period followed by a 10 seconds "off" period for total treatment time 20 minutes.
  Arms: Russian Current Stimulation + selected physical therapy exercise
Other: Placebo Russian Current Stimulation for Anterior Tibial Group — Placebo Russian current stimulation was applied to the anterior tibial group without active current for 20 minutes.
  Arms: Placebo Russian Current Stimulation + selected physical therapy exercise
Other: Selected physical therapy exercise for both limbs — The selected physical therapy exercise for both limbs was applied for 40 minutes, including passive, active assisted and active range of motion exercises, stretching of spastic muscles, strengthening of weak muscles (anterior tibial group), and finally functional mobility exercises.

SUMMARY:
This study aimed to examine the effect of Russian current stimulation on Anterior tibial group on postural stability and risk of falling in patients with stroke.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death globally and the main cause of disability, with ischemic strokes accounting for about 87% of cases. In 2010, over 11 million ischemic strokes occurred, predominantly in low and middle-income countries, leading to approximately three million deaths. Hemorrhagic strokes account for 13% of cases.

Egypt, with an estimated population of 85.5 million, has a high stroke prevalence of 963 per 100,000 inhabitants. Postural imbalance is a common limitation, affecting 83% of acute stroke patients, and falls are frequent across all stages of recovery, with rates as high as 73% within six months post-discharge. Even in chronic stroke patients, the fall risk remains elevated compared to age-matched controls. Postural imbalance impacts quality of life, and rehabilitation is vital for regaining independence in daily activities.

Up to 30% of stroke survivors experience significant permanent disabilities, and 20% require rehabilitation. Motor impairments, particularly in the lower limbs, limit daily activities, community participation, and quality of life. Poor lower-limb muscle performance affects balance, gait, and functionality, but interventions like Russian current have shown effectiveness in improving walking performance and motor recovery in chronic stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Forty patient with stroke manifest with weakness of anterior tibial group.
* Patients with moderate spasticity,
* Patient's ages ranged from 40-55 years.
* Patients BMI not exceed 30 kg/m².
* Medically and clinically stable patients.

Exclusion Criteria:

* Patients suffering from psychological, cognitive, or emotional disturbance.
* Patients with severe spasticity (3 or more by the modified Ashworth scale).
* Patients with atrial fibrillation.
* Patients with infectious processes.
* Patients with impaired pain sensitivity.
* Patients with epilepsy.
* Patients with lower limb joint endoprosthetics.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Static postural stability overall stability index (OST) | 6 weeks
  It was assessed for both groups through Biodex balance system. A training test was given to each patient followed by three consecutive tests in static mode. Each one lasted for 20 seconds with 10 seconds rest between each, changes were recorded in relation to the center of the platform, and the mean of three tests showing the postural fluctuations of women was automatically calculated by the device, and displayed on the screen of device.

SECONDARY OUTCOMES:
Berg balance scale | 6 weeks
  It was used to assess the balance for all patients in both groups. The scale consists of 14 items, scored from 0 to 4, which are added to make a total score between 0 and 56. A higher score indicates better balance. The items vary in difficulty, from sitting in a chair to standing on one leg.
Risk of falls index | 6 weeks
  Risk of falls index of all patients in both groups was assessed through Biodex balance system. All patients in both groups were asked to bilaterally stand on the locked platform; then were asked to look in front to the screen that will adjusted according to their height, the hands were placed comfortably beside the body and they were advised to use the handles of the device in case of loss of balance and repeat the test from the beginning.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Mohamed Zakaria, PhD, Study Chair — Professor, Cairo University
Locations (1):
- Deraya University, Minya, Egypt